CLINICAL TRIAL: NCT02751723
Title: Assessment of Disease Burden and Palliative Care Needs of Patients During the Course of Incurable Cancer Disease
Acronym: APM-Project
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Florian Lordick, MD (Other)
Responsible Party: Sponsor-Investigator, Florian Lordick, MD, Prof. Dr. med. (MD, PhD), University of Leipzig
Organization: University of Leipzig (Other)
Other Study IDs: APM Project; DRKS00007536 (Registry Identifier: Deutsches Register Klinischer Studien)
Record Dates: First submitted 2016-04-14; First posted 2016-04-26 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Cancer Disease, Palliative Therapy
Keywords: cancer disease; palliative care; palliative therapy; cancer; patient´s needs; patient care; disease burden
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- lung cancer: validated questionnaires
  Interventions: Other: validated questionnaires
- malignant melanoma: validated questionnaires
  Interventions: Other: validated questionnaires
- cancer of the hepatobiliary system: validated questionnaires
  Interventions: Other: validated questionnaires
- head and neck cancer: validated questionnaires
  Interventions: Other: validated questionnaires
- breast cancer: validated questionnaires
  Interventions: Other: validated questionnaires
- ovarian carcinoma: validated questionnaires
  Interventions: Other: validated questionnaires
- pancreatic cancer: validated questionnaires
  Interventions: Other: validated questionnaires
- stomach cancer: validated questionnaires
  Interventions: Other: validated questionnaires
- oesophageal cancer: validated questionnaires
  Interventions: Other: validated questionnaires
- colorectal cancer: validated questionnaires
  Interventions: Other: validated questionnaires

INTERVENTIONS:
Other: validated questionnaires

SUMMARY:
The aim of this non-investigational study is to determine the symptoms and disease burden at the time point of diagnosis and in the further course of an incurable cancer disease. The needs and preferences of patients suffering from cancer (ovarian carcinoma, breast cancer, malignant melanoma, lung cancer, stomach cancer, oesophageal cancer, pancreatic cancer, cancer of the hepatobiliary system, colorectal cancer, head and neck cancer) are examined by various validated questionnaires. The data obtained by these questionnaires are collected together with information obtained by the treating physicians at four time points during the study: t0 - patient´s enrollment, at the moment of diagnosis and before the start of tumor therapy, respectively; T1 - 3 months after patient´s enrollment; T2 - 6 months after patient´s enrollment; T3 - 12 months after patient´s enrollment. This highly innovative project offers the chance to identify medical services deficits and risk circumstances for the burden of treatments in an oncology-palliative setting and to optimize the quality of patient care.

ELIGIBILITY:
Inclusion Criteria:

* Incurable cancer disease: ovarian carcinoma, breast cancer, malignant melanoma, lung cancer, stomach cancer, oesophageal cancer, pancreatic cancer, cancer of the hepatobiliary system, colorectal cancer, head and neck cancer
* signed and dated Inform Consent Form
* Age ≥ 18 years

Exclusion Criteria:

* Patient is not able to understand and to answer questions
* Patient is in a critical health situation and is directly threatened due to cancer disease or the resulting complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with newly diagnosed incurable cancer disease before start of any tumor therapy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Patient´s answers regarding symptom burden at 12 months | 12 months after enrollment

SECONDARY OUTCOMES:
Change from Baseline physician´s report at 12 months | 12 months after enrollment
Change from Baseline Patient´s answers regarding symptom burden at 6 months | 6 months after enrollment
Change from Baseline physician´s report at 6 months | 6 months after enrollment
Change from Baseline Patient´s answers regarding symptom burden at 3 months | 3 months after enrollment
Change from Baseline physician´s report at 3 months | 3 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Florian Lordick, Prof. Dr., Study Chair — University of Leipzig; Bend Alt-Epping, PD Dr., Study Chair — University of Göttingen; Anja Mehnert, Prof. Dr., Study Chair — University of Leipzig; Birgitt van Oorschot, Prof. Dr., Study Chair — Comprehensive Cancer Centre Main-Franken, Würzburg; Michael Thomas, Prof. Dr., Study Chair — Heidelberg University
Locations (21):
- Germany (21):
  - UCCL, University of Leipzig, Leipzig, Saxony
  - Municipal Hospital Braunschweig, Braunschweig
  - Internal medicine practice, Burgwedel
  - Municipal Hospital Essen-Mitte, Essen
  - University of Essen, Essen
  - University of Göttingen, Göttingen
  - University of Hamburg-Eppendorf, Hamburg
  - Medical University Hanover, Hanover
  - Clinic for Thoraric Diseases (Thoraxklinik), Heidelberg
  - Municipal Hospital Karlsruhe, Karlsruhe
  - University of Leipzig, ENT, Leipzig
  - Hospital Leverkusen, Leverkusen
  - Municipal Hospital Magdeburg, Magdeburg
  - University of Mainz, Mainz
  - Maria Hilf Clinic, Mönchengladbach
  - Radiotherapy practice, Recklinghausen
  - University of Regensburg, Regensburg
  - Hospital Südstadt Rostock, Rostock
  - Immanuel Hospital Rüdersdorf, Rüdersdorf
  - Hospital Traunstein, Traunstein
  - Comprehensive Cancer Centre Main-Franken, Würzburg

IPD SHARING:
Plan to Share IPD: No